CLINICAL TRIAL: NCT02856802
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Efficacy and Safety Study of DFN-02 in Episodic Migraine With or Without Aura
Brief Title: An Efficacy and Safety Study of DFN-02 (Sumatriptan Nasal Spray 10 mg)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Upsher-Smith Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DFN-02-CD-012
Record Dates: First submitted 2016-07-29; First posted 2016-08-05 (Estimated); Results first posted 2021-03-30 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2020-12

CONDITIONS: Migraine Headaches
Keywords: Aura
MeSH Terms: conditions — Migraine Disorders; Epilepsy | interventions — Sumatriptan; Nasal Sprays

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DFN-02 (Experimental): Participants self-administered a single-dose of DFN-02 (sumatriptan 10-mg/100 μL nasal spray) intranasally within one hour of an acute migraine pain episode.
  Interventions: Drug: Sumatriptan 10 mg Nasal Spray
- Placebo (Other): Participants self-administered a single-dose of DFN-02 placebo nasal spray matching DFN-02 intranasally within one hour of an acute migraine pain episode.
  Interventions: Other: Sumatriptan Placebo Nasal Spray

INTERVENTIONS:
Drug: Sumatriptan 10 mg Nasal Spray — 100 μL nasal spray once
  Other Names: Sumatriptan
  Arms: DFN-02
Other: Sumatriptan Placebo Nasal Spray — 100 μL nasal spray once
  Arms: Placebo

SUMMARY:
A safety and efficacy study of DFN-02 (Sumatriptan Nasal Spray 10 mg), being conducted at multiple centers in the United States.

DETAILED DESCRIPTION:
This was a randomized, two double-blind (DB) treatment period dosing study.

Previously diagnosed subjects with a history of episodic migraine (as defined by International Classification of Headache Disorders (ICHD), 3rd edition [beta version] [ICHD 3]) who experienced an average of 2 to 8 migraine attacks per month for at least the prior 12 months, with no more than 14 headache days per month, and with 48 hours of headache free time between migraine, were randomized in a 1:1 ratio in both DB periods to receive either DFN-02 (sumatriptan nasal spray 10 mg) or a matching placebo.

Subjects treated one moderate to severe migraine attack in the first double-blind treatment period (DB1) and, if eligible, were re-randomized into the second double-blind treatment period (DB2) to treat another migraine attack at any pain level.

There was a screening period of up to 21 days to evaluate whether subjects fit the migraine inclusion criteria pursuant to ICHD-3, and did not have medication overuse. Subjects with at least a 12 month medical history of acute migraine were eligible for enrollment in the treatment period. Subjects continued to take their normal migraine medication during this screening period.

If eligible and randomized, subjects in the DB1 treatment period were instructed to use the study medication in one migraine attack as soon as (and no more than within one hour after) experiencing moderate to severe migraine pain (defined as headache pain rating of Grade 2 [moderate] or Grade 3 [severe] on a pain severity scale of 0 to 3). If the subject was not able to use study medication for the first migraine after randomization, they were instructed to use the study medication for the next attack. Those subjects who did not experience a migraine attack, and/or did not treat any migraine attack with study medication or record diary data, were not allowed to continue into the DB2 treatment period, and were discontinued.

After treating a migraine attack with study medication, subjects were instructed to contact the site within 24 hours of the treated migraine (or the next working day) to schedule their next visit.

Subjects returned to the study site within 2 to 7 days in the DB1 treatment period and, if continuing to be eligible, were re-randomized into a DB2 treatment period to treat one migraine attack at any pain level, and return to the study site within 2 to 7 days of the second treatment.

Once randomized, the total duration of each subject's participation in the study was up to 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. A history of episodic migraine who experience an average of 2 to 8 migraine attacks per month for at least the past 12 months, with no more than 14 headache days per month, and with 48 hours of headache free time between migraine headaches
2. Patients who have migraine with or without aura. If migraine with aura, the aura cannot last longer than 60 minutes.
3. Patients who are willing and able to:

   1. Evaluate and record pain, migraine symptoms, and study medication effectiveness information in real-time using a diary for the duration of the study;
   2. Record each instance of the use of study medication and rescue medication in a patient diary in real-time for the duration of the study;
   3. Comply with all other study procedures and scheduling requirements.

Exclusion Criteria:

1. Minors, even if they are in the specified study age range
2. Medication overuse:

   1. Opioids ≥ 10 days during the 90 days prior to screening
   2. Combination medications (e.g., Fiorinal®) ≥ 10 days during the 90 days prior to screening (only applies if combination medication contains an opioid and/or barbiturate)
   3. Nonsteroidal Anti-inflammatory Drugs or other simple medications ˃ 14 days a month during the 90 days prior to screening
   4. Triptans or ergots ≥ 10 days a month during the 90 days prior to screening
3. Treated with onabotulinumtoxinA (Botox®) or other botulinum toxin treatment within 4 months prior to screening for migraine prophylaxis (patients who were treated with same for cosmetic purposes may be allowed on a case-by-case basis after approval from the Medical Monitor)
4. A history of or current neurological or psychiatric impairment, or cognitive dysfunction that, in the opinion of the Investigator, would compromise data collection
5. Use of antipsychotics at least 15 days prior to randomization
6. Patients who received treatment with an investigational drug or device within 30 days prior to randomization, or within 3 months if associated with central nervous system
7. Patients who participated in a central nervous system clinical trial within 3 months prior to randomization
8. Patients who test positive for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) antibody serology testing
9. Patients who are employees or immediate relatives of the employees of the Sponsor, any of its affiliates or partners, or of the clinical study research site

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2016-07-11 (Actual); Primary Completion 2017-02-10 (Actual); Study Completion 2017-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sagar Munjal, MD, Study Director — Dr. Reddy's Laboratories, LLC
Locations (9):
- United States (9):
  - Site 30, San Diego, California
  - Site 11, Santa Monica, California
  - Site 31, Boston, Massachusetts
  - Site 18, Ann Arbor, Michigan
  - Site 02, Albuquerque, New Mexico
  - Site 29, Rochester, New York
  - Site 25, Williamsville, New York
  - Site 33, Mt. Pleasant, South Carolina
  - Site 28, West Jordan, Utah

REFERENCES:
- [Derived] Lipton RB, Munjal S, Brand-Schieber E, Rapoport AM. DFN-02, Sumatriptan 10 mg Nasal Spray with Permeation Enhancer, for the Acute Treatment of Migraine: A Randomized, Double-Blind, Placebo-Controlled Study Assessing Functional Disability and Subject Satisfaction with Treatment. CNS Drugs. 2019 Apr;33(4):375-382. doi: 10.1007/s40263-019-00614-6. PMID 30877622
- [Derived] Lipton RB, Munjal S, Brand-Schieber E, Rapoport AM. DFN-02 (Sumatriptan 10 mg With a Permeation Enhancer) Nasal Spray vs Placebo in the Acute Treatment of Migraine: A Double-Blind, Placebo-Controlled Study. Headache. 2018 May;58(5):676-687. doi: 10.1111/head.13309. PMID 29878341

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in the United States. At least 1 subject was enrolled at 9 study centers.
Pre-assignment Details: Subjects had to have an average of 2 to 8 migraine attacks per month for at least the prior 12 months, with no more than 14 headache days per month, and with 48 hours of headache free time between migraine.
Groups:
- DFN-02: DFN-02 Active Nasal Sumatriptan 10mg spray upon onset of acute migraine pain during each acute migraine episode
  DFN-02
- Placebo: DFN-02 Placebo spray upon onset of acute migraine pain during each acute migraine episode
  DFN-02 Placebo
Period: Double-Blind Treatment Period 1
Arm/Group | DFN-02 | Placebo
Started | 50 (4 of 54 randomized subjects did not start; 2 had no migraines, 1 withdrew, 1 lost to follow-up.) | 43 (10 of 53 randomized subjects did not start; 6 had no migraines, 3 withdrew, 1 sponsor terminated.)
Completed | 48 | 38
Not Completed | 2 | 5
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Sponsor terminated | 1 | 0
Not completed — Lack of diary compliance | 0 | 2
Period: Double-Blind Treatment Period 2
Arm/Group | DFN-02 | Placebo
Started (86 subjects completing double-blind treatment period 1, and still eligible, were re-randomized into double-blind treatment period 2) | 37 (6 of 43 re-randomized subjects did not start; 5 had no migraines, for 1 protocol deviation.) | 38 (5 of 43 re-randomized subjects did not start; 4 had no migraines, for 1 prohibited drug use.)
Completed | 36 | 38
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: A maximum 21 day screening period was conducted to evaluate whether a subject met the migraine inclusion criteria pursuant to ICHD-3, and did not exhibit medication overuse. If eligible and randomized, subjects in the DB1 treatment period were instructed to use the study medication for their first migraine attack as soon as (and no more than 1 hour after) experiencing moderate to severe migraine pain. If the subject was missed dosing the first migraine, they were to dose the next attack.
Groups:
- DFN-02 (Double-Blind Treatment Period 1): 50 of 54 randomized subjects started and were dosed; 2 subjects had no migraine attack, 1 subject withdrew and 1 subject was lost to follow-up. Per protocol these 4 subjects are excluded from analysis.
- Placebo (Double-Blind Treatment Period 1): 43 of 53 randomized subjects started and were dosed; 6 subjects had no migraine attack, 3 subjects withdrew and 1 subject was terminated by the sponsor. Per protocol these 10 subjects are excluded from analysis.
- Total: Total of all reporting groups
Arm/Group | DFN-02 (Double-Blind Treatment Period 1) | Placebo (Double-Blind Treatment Period 1) | Total
Number analyzed (Participants) | 50 | 43 | 93
Age, Continuous [Mean (Full Range); unit: years] | 43.4 [20 to 68] | 41.0 [19 to 63] | 42.3 [19 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 37 | 75
  Male | 12 | 6 | 18
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 0 | 1 | 1
  Black or African American | 5 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  White | 42 | 40 | 82
  Other | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 50 | 43 | 93
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.70 (6.441) | 28.80 (7.500) | 28.21 (6.933)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Free From Headache Pain at 2 Hours After the First Dose of Study Medication Taken for a Migraine Attack With Moderate to Severe Headache Pain During the Double-blind Treatment Period 1 (DB1).
Description: Freedom from headache pain at 2 hours after the first dose of study medication taken within one hour after experiencing a migraine attack of moderate to severe headache pain during the DB1 treatment period, e.g., headache pain rating of moderate [Grade 2] or severe [Grade 3] predose and reduced to none [Grade 0] postdose). Mild headache pain was recorded as Grade 1. If the subject was not able to use study medication for the first migraine after randomization, they were instructed to use the study medication for the next attack. If the subject experienced insufficient relief from the first dose of study medication, they were permitted to take a second dose of study medication or rescue medication 2 or more hours after the first dose, and only after completing the 2 hours' postdose assessments. If no relief was experienced from the first dose of study medication after 2 hours only rescue medication could be administered. Maximum 2 doses of study medication per 24 hours.
Time Frame: 2 hours after study medication administration
Population: Full Analysis Set (FAS) population. Last observation carried forward (LOCF) imputation method. The FAS included all randomized subjects who took at least one dose of study medication during the DB treatment period (1) and had at least one post-baseline efficacy time point assessment in DB treatment period (1).
Measure: Count of Participants; unit: Participants
Groups:
- DFN-02 (DB1): DFN-02 Active Nasal Sumatriptan 10mg spray upon onset of acute migraine pain during each acute migraine episode
  DFN-02
- Placebo (DB1): DFN-02 Placebo spray upon onset of acute migraine pain during each acute migraine episode
  DFN-02 Placebo
Arm/Group | DFN-02 (DB1) | Placebo (DB1)
Number analyzed (Participants) | 48 | 40
Participants | 21 | 9
Statistical Analysis 1: Comparison: DFN-02 (DB1) vs Placebo (DB1); Statistical testing and confidence intervals (CIs) were 2 sided and performed using a significance (alpha) level of 0.05. All statistical analyses were conducted with the statistical analysis system (SAS)® software package (version 9.3); Test type: Non-Inferiority — Assumption that 15% of placebo and 42% of DFN 02 10 mg (treated) subjects would be pain-free at 2 hours. A sample size of 50 subjects in each DB1 dosing arm provided 86% power to detect this assumed difference between placebo and DFN-02 10 mg at a 5% (2-sided) level of significance; p = 0.044, Fisher Exact; Odds Ratio (OR) = 2.68, 95% CI 2-sided [1.05 to 6.83]

2. Secondary Outcome: Number of Participants With Absence of Most Bothersome Symptom (MBS) Among Nausea, Photophobia and Phonophobia at 2 Hours (DB1)
Description: Number of participants with their MBS among nausea, photophobia and phonophobia absent at 10, 15, 20, 30, 60, 90, and 120 minutes after the first dose of study medication taken for a migraine attack during DB1 treatment period are summarized by treatment group and time point for the full analysis set (FAS1). The corresponding p-values from Fisher's exact test were computed for the comparison between treatment groups. Subjects who reported a MBS predose and reported the status of the MBS at the particular postdose time point were analyzed.
Time Frame: 2 hours after study medication administration
Population: Subjects who reported a MBS predose and reported the status of the MBS at the particular postdose time point were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | DFN-02 (DB1) | Placebo (DB1)
Number analyzed (Participants) | 41 | 38
Participants | 29 | 15
Statistical Analysis 1: Comparison: DFN-02 (DB1) vs Placebo (DB1); Test type: Non-Inferiority — Non-inferiority conducted as specified in the statistical analysis plan (SAP); p = 0.007, Fisher Exact — The corresponding p-values from Fisher's exact test were computed for the comparison between treatment groups

3. Secondary Outcome: Number of Participants With Headache Pain Freedom at 2 Hours Postdose in the Double-blind Treatment Period 2 (DB2)
Description: In Double-blind Treatment Period 2 (DB2), freedom from headache pain 2 hours after the first dose of study medication taken within one hour of experiencing a migraine attack for any headache pain level, e.g., mild [Grade 1], moderate [Grade 2], or severe [Grade 3] and reduced to none [Grade 0] after study medication administration. If the subject was not able to use study medication for the first migraine after randomization, they were instructed to use the study medication for the next attack.
Time Frame: 2 hours after study medication administration
Population: Last observation carried forward (LOCF) imputation method. Analysis included all randomized subjects who took at least one dose of study medication during the second DB treatment period (2) and had at least one post-baseline efficacy time point assessment in DB treatment period (2).
Measure: Count of Participants; unit: Participants
Groups:
- DFN-02 (DB2): Participants self-administered a single-dose of DFN-02 (sumatriptan 10-mg/100 μL nasal spray) intranasally within one hour of an acute migraine pain episode.
  Sumatriptan 10 MG Nasal Spray: 100 μL nasal spray once
- Placebo (DB2): Participants self-administered a single-dose of DFN-02 placebo nasal spray matching DFN-02 intranasally within one hour of an acute migraine pain episode.
  Sumatriptan Placebo Nasal Spray: 100 μL nasal spray once
Arm/Group | DFN-02 (DB2) | Placebo (DB2)
Number analyzed (Participants) | 36 | 37
Participants | 19 | 17
Statistical Analysis 1: Comparison: DFN-02 (DB2) vs Placebo (DB2); Statistical testing and confidence intervals (CIs) were 2 sided and performed using a significance (alpha) level of 0.05. All statistical analyses were conducted with the SAS® software package (version 9.3); Test type: Non-Inferiority — No assumptions made; p = 0.642, Fisher Exact; Odds Ratio (OR) = 1.31, 95% CI 2-sided [0.52 to 3.30]

ADVERSE EVENTS:
Time Frame: Adverse Events were assessed from the initial dose of study medication up to 5 days after the last dose of study medication.
Groups:
- DFN-02 (DB1): DFN-02 Active Nasal Sumatriptan 10-mg spray upon onset of acute migraine pain during each acute migraine episode
  DFN-02 Active in Double-blind Treatment Period 1
- Placebo (DB1): DFN-02 Placebo spray upon onset of acute migraine pain during each acute migraine episode
  DFN-02 Placebo in Double-blind Treatment Period 1
- DFN-02 (DB2): DFN-02 Active Nasal Sumatriptan 10-mg spray upon onset of acute migraine pain during each acute migraine episode
  DFN-02 Active in Double-blind Treatment Period 2
- Placebo (DB2): DFN-02 Placebo spray upon onset of acute migraine pain during each acute migraine episode
  DFN-02 Placebo in Double-blind Treatment Period 2
Arm/Group | DFN-02 (DB1) | Placebo (DB1) | DFN-02 (DB2) | Placebo (DB2)
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/43 | 0/37 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/43 | 0/37 | 0/38
Other Adverse Events (participants affected / at risk) | 5/50 | 0/43 | 5/37 | 0/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DFN-02 (DB1) (N=50) | Placebo (DB1) (N=43) | DFN-02 (DB2) (N=37) | Placebo (DB2) (N=38)
Application site pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Chest Discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Burning sensation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-06-01): https://cdn.clinicaltrials.gov/large-docs/02/NCT02856802/Prot_000.pdf
  • Statistical Analysis Plan (2016-09-16): https://cdn.clinicaltrials.gov/large-docs/02/NCT02856802/SAP_001.pdf